CLINICAL TRIAL: NCT05781529
Title: Injectable Platelets Rich Fibrin Versus Hyaluronic Acid With Bovine Derived Xenograft for Alveolar Ridge Preservation (A Randomized Controlled Clinical Trial With Histomorphometric Analysis)
Brief Title: Injectable Platelets Rich Fibrin Versus Hyaluronic Acid for Alveolar Ridge Preservation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21832
Record Dates: First submitted 2023-02-28; First posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Alveolar Ridge Enlargement
MeSH Terms: interventions — Alveolar Ridge Augmentation; Hyaluronic Acid; Transplantation, Heterologous

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Injectable platelets rich fibrin (Experimental): Injectable platelets rich fibrin was prepared where 10 ml of patient venous blood was centrifuged without anti-coagulants (plain plastic glass-coated) at 700 rpm speed for only 3 minutes, xenograft was mixed with I-PRF to make sticky bone, sticky bone was placed into extraction socket till the socket was fully filled up to the gingival margin
  Interventions: Procedure: Alveolar ridge augmentation with injectable platelets rich fibrin
- Hyaluronic acid (Experimental): Hyaluronic acid (HA) syringe containing 1 mL of cross-linked hyaluronic at a concentration of 20 mg/ml in a saline phosphate buffer solution at sterilized content was used. HA was mixed with particulate xenograft 1:10 ratio to form a putty consistency for condensation and was placed into extraction socket till the socket was fully filled up to the gingival margin
  Interventions: Procedure: Alveolar ridge augmentation with hyaluronic acid
- Xenograft (Active Comparator): Xenograft was mixed with saline, placed in extraction socket till the socket is fully filled up to the gingival margin
  Interventions: Procedure: Alveolar ridge augmentation with xenograft

INTERVENTIONS:
Procedure: Alveolar ridge augmentation with injectable platelets rich fibrin — Injectable platelets rich fibrin is added to xenograft for alveolar ridge augmentation in order to preserve bone and decrease bone resorption
  Other Names: Socket augmentation with injectable platelets rich fibrin
  Arms: Injectable platelets rich fibrin
Procedure: Alveolar ridge augmentation with hyaluronic acid — Hyaluronic is added to xenograft for alveolar ridge augmentation in order to preserve bone and decrease bone resorption
  Other Names: Socket augmentation with hyaluronic acid
  Arms: Hyaluronic acid
Procedure: Alveolar ridge augmentation with xenograft — Xenograft is added alone as a active compatator
  Other Names: Socket augmentation with xenograft
  Arms: Xenograft

SUMMARY:
Thirty-six patients (19 females and 17 males) that required implant placement in esthetic zone participated in this study and were blindly allocated 12 patients per group, all patients had ARP either with I-PRF with xenograft, HA with xenograft or xenograft alone, the sockets were sealed with free gingival graft harvested from the palate.

DETAILED DESCRIPTION:
The aim of this study was to compare injectable platelets rich fibrin (I-PRF) versus hyaluronic acid (HA) in combination with xenografts for ARP. Methods: Thirty-six patients (19 females and 17 males) that required implant placement in esthetic zone participated in this study and were blindly allocated 12 patients per group, all patients had ARP either with I-PRF with xenograft, HA with xenograft or xenograft alone, the sockets were sealed with free gingival graft harvested from the palate. The assessment was done by cone beam CT preoperative and 4 months postoperative to assess radiographic bone gain and crestal bone loss. Clinical parameters were soft tissue thickness, keratinized gingiva and clinical bone width that were assessed preoperative, 4 months and 1 year postoperative. Histological assessment of core bone biopsies 4 months postoperatively was performed by histomorphometric analysis of newly formed bone %, mature bone% and residual graft%

ELIGIBILITY:
Inclusion Criteria:

* non-restorable tooth located in anterior maxillary arch (upper right second premolar to upper left second premolar)
* socket type I according to Elian et al., 2007 classification
* tooth to be extracted was free from acute periapical infection or sinus tracts
* thick gingival biotype
* Systemically free according to modified Cornell medical index

Exclusion Criteria:

* smokers patients
* bruxism habits
* patients with poor oral hygiene or not willing to perform oral hygiene measures

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Radiographic bone width | 4 months postoperative
  Cone beam CT (CBCT) were obtained preoperatively and 4 months postoperatively. The radiographs were analyzed using One- Viewer viewing software (iCATVision). The buccolingual width was measured into different levels. At the bone crest (A), 3mm from the bone crest (B) and 6 mm from the bone crest (C). For standardization in the sagittal slice, the axial plane was adjusted to pass through the cemento enamel junction (CEJ) of the adjacent teeth. On the axial slice, the mesiodistal dimension from the distal surface to mesial surface of the adjeceent teeth was measured. The coronal plane was adjusted to be pass through the middle of the distance in order to be perpendicular to both buccal and lingual cortices. Measurement were all performed on the coronal slices. In addition, fusion was done by superimposing preoperative and 4 months CBCT in all groups.

SECONDARY OUTCOMES:
histological and histomorphometric assessment | 4 months postoperative
  The biopsy samples were harvested and processed. All samples were serially sectioned using a microtome. Slides were stained separately with hematoxylin and eosin and observed using a light microscope. For histological evaluation and histomorphometric analysis, 20 photomicrographs from different sections taken at every 200 µm of each biopsy sample were captured at original magnification 10×, 20×, and 40× using a digital camera. The image analyzer was calibrated to automatically convert the measurement units (pixels) produced by the image analyzer program into actual micrometer units. Data from the sections of each group were averaged.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Doaa Adel Salah Khattab, Cairo, Abbassia
  - Doaa Khattab, Cairo, Abbassia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Abaza G, Abdel Gaber HK, Afifi NS, Adel-Khattab D. Injectable platelet rich fibrin versus hyaluronic acid with bovine derived xenograft for alveolar ridge preservation. A randomized controlled clinical trial with histomorphometric analysis. Clin Implant Dent Relat Res. 2024 Feb;26(1):88-102. doi: 10.1111/cid.13289. Epub 2023 Oct 31. PMID 37905704